CLINICAL TRIAL: NCT00414492
Title: Pattern of Cell Death Following Neoadjuvant Therapy for Metastatic Colon Cancer
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Michael Choti, M.D., Johns Hopkins University
Other Study IDs: J06106; NA_00004883
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; liver metastasis; tumor margins; neoadjuvant therapy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — liver tissue from surgical specimen

SUMMARY:
Systemic chemotherapy for metastatic colon cancer is often used in the neoadjuvant setting for patients undergoing liver resection. This treatment is given either to keep the tumor at bay or reduce its size before the time of resection. While many metastatic tumors might appear to respond well and even radiographically disappear following neoadjuvant therapy, it is unclear whether grossly or radiographically negative areas of previous disease are microscopically free of tumor cells. As such, when possible, resection boarders typically follow 1 cm margins from the tumor size prior to neoadjuvant therapy. These margins might be necessary to encompass all histologically present disease or they might be unnecessarily large, serving only to increase the mortality and morbidity of the operation. This study begins to address this question by a histological examination of the pattern of cell death in areas of metastases removed after neoadjuvant therapy. Furthermore, clinical cases in which neoadjuvant therapy allowed for resection of previously unresectable cancer will be examined to determine whether there is an increased rate of recurrence despite "negative" resection boundaries in these cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years old.
* Patients must have colon cancer metastases to the liver.
* Patients must be candidates and be scheduled for liver resection.
* Patients must have received and have had a response to neoadjuvant therapy prior to liver resection.
* Patients must have signed Institutional Review Board (IRB) approved written consent form prior to registering in the study.

Exclusion Criteria:

* Patients who are < 18 years old.
* Patients who do not have colon cancer metastases to the liver.
* Patients who are not surgical candidates.
* Patients who do not schedule or who cancel a liver resection.
* Patients who have not received neoadjuvant therapy.
* Patients who have received neoadjuvant therapy but who have had no response or who have had tumor progression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer metastases to the liver
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-12; Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Choti, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medicine, Baltimore, Maryland, United States